CLINICAL TRIAL: NCT02350309
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Way Crossover Study to Evaluate the Effect of 2 Dosage Strengths of E2006 on a Multiple Sleep Latency Test in Subjects With Insomnia Disorder
Brief Title: Study to Evaluate the Effect of 2 Dosage Strengths of Lemborexant (E2006) on a Multiple Sleep Latency Test in Participants With Insomnia Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E2006-A001-107
Record Dates: First submitted 2015-01-07; First posted 2015-01-29 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2016-12

CONDITIONS: Insomnia Disorder
Keywords: Insomnia Disorder; E2006; Multiple Sleep Latency Test; Lemborexant
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant; Flurazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- Lemborexant 5 mg (Experimental): Participants will receive a single, oral tablet formulation dose of lemborexant 5 mg within 5 minutes before bedtime.
  Interventions: Drug: Lemborexant 5 mg
- Lemborexant 10 mg (Experimental): Participants will receive a single, oral tablet formulation dose of lemborexant 10 mg within 5 minutes before bedtime.
  Interventions: Drug: Lemborexant 10 mg
- Lemborexant-matched Placebo (Placebo Comparator): Participants will receive a single, oral tablet formulation dose of lemborexant-matched placebo within 5 minutes before bedtime.
  Interventions: Drug: Lemborexant-matched placebo.
- Flurazepam 30 mg (Active Comparator): Participants will receive a single, oral capsule formulation dose of flurazepam 30 mg within 5 minutes before bedtime.
  Interventions: Drug: Flurazepam 30 mg

INTERVENTIONS:
Drug: Lemborexant 5 mg — Lemborexant 5 mg tablet.
  Other Names: E2006
  Arms: Lemborexant 5 mg
Drug: Lemborexant 10 mg — Lemborexant 10 mg tablet.
  Other Names: E2006
  Arms: Lemborexant 10 mg
Drug: Lemborexant-matched placebo. — Lemborexant-matched placebo tablet.
  Other Names: E2006
  Arms: Lemborexant-matched Placebo
Drug: Flurazepam 30 mg — Flurazepam 30 mg capsule.
  Arms: Flurazepam 30 mg

SUMMARY:
This is a single-dose, randomized, placebo-controlled, 3-way crossover study of 2 dosage strengths of lemborexant (5 mg and 10 mg) in participants with insomnia disorder.

DETAILED DESCRIPTION:
The study will have 2 phases: Prerandomization and Randomization. The Prerandomization Phase will consist of 2 periods that taken together, will last up to a maximum of 21 days: a Screening Period and a Baseline Period. The Randomization Phase will comprise 4 treatment periods (Treatment 1, Treatment 2, Treatment 3, Treatment 4) with intervening washout periods between treatment periods (Washout 1, Washout 2, Washout 3). A single dose of study drug will be administered in a randomized, 3-way double-blind crossover manner at Treatment Periods 1-3; flurazepam 30 mg will be administered in an open-label manner at Treatment Period 4.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 or older, at the time of informed consent.
2. Meets the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for Insomnia Disorder, as follows:

   1. Complains of dissatisfaction with nighttime sleep despite adequate opportunity for sleep, with complaint being one or more of the following: difficulty getting to sleep, difficulty staying asleep, or awakening earlier in the morning than desired.
   2. Frequency of complaint greater than or equal to 3 times per week.
   3. Duration of complaint greater than or equal to 3 months.
   4. Associated with complaint of daytime impairment.
3. Insomnia Severity Index score greater than or equal to 15 at Screening.
4. Regular time in bed between 7 and 9 hours as reported at Screening.
5. Regular bedtime, defined as the time the participant attempts to fall asleep, between 21:00 and 24:00 and regular wake time between 05:00 and 09:00 as reported at Screening.
6. Confirmation of current insomnia symptoms as determined from responses on the Sleep Diary completed for 7 nights during Screening, such that participant Sleep Onset Latency (sSOL) greater than or equal to 30 minutes on at least 3 nights and subjective Wake After Sleep Onset (sWASO) greater than or equal to 60 minutes on at least 3 nights.

Exclusion Criteria:

1. Excessive morning sleepiness at Baseline as determined by average SOL at Baseline less than 10 minutes.
2. Females must not be lactating or pregnant at Screening or Baseline (documented by a negative beta-human chorionic gonadotropin [beta-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of beta-hCG or hCG). (Note: A negative urine pregnancy test is required at check-in before each dose of study drug and flurazepam).
3. If females of childbearing potential:

   1. Had unprotected sexual intercourse within 30 days before study entry and do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation.
   2. Are currently abstinent, and do not agree to use a double barrier method (as described above) or refrain from sexual activity during the study period or for 28 days after study drug discontinuation.
   3. Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation.

   NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
4. A current diagnosis of sleep-related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or narcolepsy, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia.
5. Reports experiencing within the past year confusional arousals, symptoms of REM Behavior Disorder, or sleep-related violent behavior on Munich Parasomnia Scale (MUPS), or a history of aberrant nocturnal behaviors including sleep-driving or sleep-eating.
6. Habitually naps more than 3 times per week.
7. History of drug or alcohol dependency or abuse within approximately the last 2 years.
8. Has a positive drug screen at Screening.
9. A prolonged QT/QTc interval (QTc greater than 450 ms) as demonstrated by a repeated ECG at Screening (repeated only if initial ECG indicates a QTc interval greater than 450 ms).
10. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening or any lifetime suicidal behavior.
11. Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, renal, psychiatric or neurological disease, or chronic pain) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments.
12. Used any prohibited prescription or over-the-counter concomitant medications within 2 weeks prior to Screening, or between Screening and Randomization.
13. Used any modality of treatment for insomnia, including cognitive behavioral therapy or marijuana within 2 weeks prior to Screening, or between Screening and Randomization.
14. Scheduled for surgery during the study.
15. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Baseline, or plans to travel more than 3 times zones during the study.
16. Hypersensitivity to flurazepam, the study drug, or any of the excipients.
17. Currently enrolled in another clinical trial or used any investigational drug or device within 28 days or 5 x the half-life, whichever is longer preceding informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-12-13 (Actual); Primary Completion 2015-04-21 (Actual); Study Completion 2015-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atlanta, Georgia
  - Crestview Hills, Kentucky

REFERENCES:
- [Derived] Mayleben D, Rosenberg R, Pinner K, Hussein Z, Moline M. Assessment of morning sleep propensity with lemborexant in adults with insomnia disorder in a randomized, placebo-controlled crossover study. Sleep Adv. 2021 Jul 2;2(1):zpab011. doi: 10.1093/sleepadvances/zpab011. eCollection 2021. PMID 37193566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United Sates from 13 December 2014 to 21 April 2015.
Pre-assignment Details: A total of 123 participants were screened, of which 54 participants were screen failures and 69 participants were randomized to receive study treatment.
Groups:
- Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg: Participants received a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Period 1, followed by a single oral dose of lemborexant 5 milligrams (mg) tablet, on Day 1 of Treatment Period 2, followed by a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Period 3, followed by a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4. All doses were administered within 5 minutes before bedtime. A washout period of 12 to 16 days was maintained between the 2 treatment periods.
- Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg: Participants received a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Period 1, followed by a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Period 2, followed by a single oral dose of lemborexant 5 mg tablet, on Day 1 of Treatment Period 3, followed by a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4. All doses were administered within 5 minutes before bedtime. A washout period of 12 to 16 days was maintained between the 2 treatment periods.
- Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg: Participants received a single oral dose of lemborexant 5 mg tablet, on Day 1 of Treatment Period 1, followed by a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Period 2, followed by a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Period 3, followed by a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4. All doses were administered within 5 minutes before bedtime. A washout period of 12 to 16 days was maintained between the 2 treatment periods.
- Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg: Participants received a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Period 1, followed by a single oral dose of lemborexant 5 mg tablet, on Day 1 of Treatment Period 2, followed by a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Period 3, followed by a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4. All doses were administered within 5 minutes before bedtime. A washout period of 12 to 16 days was maintained between the 2 treatment periods.
- Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg: Participants received a single oral dose of lemborexant 5 mg tablet, on Day 1 of Treatment Period 1, followed by a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Period 2, followed by a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Period 3, followed by a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4. All doses were administered within 5 minutes before bedtime. A washout period of 12 to 16 days was maintained between the 2 treatment periods.
- Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg: Participants received a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Period 1, followed by a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Period 2, followed by a single oral dose of lemborexant 5 mg tablet, on Day 1 of Treatment Period 3, followed by a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4. All doses were administered within 5 minutes before bedtime. A washout period of 12 to 16 days was maintained between the 2 treatment periods.
Period: Treatment Period 1 (2 Days)
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg
Started | 12 | 11 | 11 | 11 | 12 | 12
Completed | 12 | 11 | 10 | 11 | 12 | 12
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period 1 (12-16 Days)
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg
Started | 12 | 11 | 10 | 11 | 12 | 12
Completed | 12 | 11 | 10 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (2 Days)
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg
Started | 12 | 11 | 10 | 11 | 12 | 12
Completed | 12 | 11 | 10 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (12-16 Days)
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg
Started | 12 | 11 | 10 | 11 | 12 | 12
Completed | 12 | 11 | 10 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (2 Days)
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg
Started | 12 | 11 | 10 | 11 | 12 | 12
Completed | 12 | 11 | 10 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (12-16 Days)
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg
Started | 12 | 11 | 10 | 11 | 12 | 12
Completed | 12 | 11 | 10 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4 (2 Days)
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg
Started | 12 | 11 | 10 | 11 | 12 | 12
Completed | 12 | 11 | 10 | 11 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death in the Family | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of participants who received at least one dose of study drug and had at least 1 postdose safety assessment.
Groups:
- Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg: Participants received a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Period 1, followed by a single oral dose of lemborexant 5 mg tablet, on Day 1 of Treatment Period 2, followed by a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Period 3, followed by a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4. All doses were administered within 5 minutes before bedtime. A washout period of 12 to 16 days was maintained between the 2 treatment periods.
- Total: Total of all reporting groups
Arm/Group | Placebo, Lemborexant 5 mg, Lemborexant 10 mg, Flurazepam 30 mg | Lemborexant 10 mg, Placebo, Lemborexant 5 mg, Flurazepam 30 mg | Lemborexant 5 mg, Lemborexant 10 mg, Placebo, Flurazepam 30 mg | Lemborexant 10 mg, Lemborexant 5 mg, Placebo, Flurazepam 30 mg | Lemborexant 5 mg, Placebo, Lemborexant 10 mg, Flurazepam 30 mg | Placebo, Lemborexant 10 mg, Lemborexant 5 mg, Flurazepam 30 mg | Total
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 12 | 12 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (15.73) | 50.2 (12.54) | 49.0 (12.32) | 52.5 (15.91) | 48.1 (13.90) | 52.2 (7.86) | 50.2 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 10 | 9 | 7 | 8 | 51
  Male | 3 | 3 | 1 | 2 | 5 | 4 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 11 | 11 | 12 | 12 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 7 | 3 | 6 | 5 | 33
  White | 7 | 4 | 4 | 8 | 5 | 7 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Average Sleep Onset Latency (SOL) From Modified-Multiple Sleep Latency Test (M-MSLT) for Each Treatment in Treatment Periods 1 to 3
Description: SOL is defined as the length of time that it takes to accomplish the transition from full wakefulness to sleep. The multiple sleep latency test (MSLT) is a widely used method for objectively quantifying excessive, pathological, or pharmacologically induced residual sleepiness by measuring the number of minutes that it takes a participant to fall asleep. The MSLT was modified to include four Sleep Latency Tests (SLTs), with the first starting at 45 minutes after morning wake time, and the subsequent three occurring at 30-minute intervals for a total of 4 SLT's per M-MSLT. Each SLT was scored to determine the latency in minutes (with precision to 0.5 minute) from lights off to sleep onset; trials during which sleep onset did not occur were assigned a latency of 20 minutes. The four SLTs for each participant were averaged to obtain the mean SOL.
Time Frame: Baseline, Day 2 of each of three treatment periods that were separated by approximately 2 weeks (for a total of up to 4 weeks)
Population: The full analysis set (FAS) was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose pharmacodynamics (PD) measurement.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Lemborexant-matched Placebo: Participants received a single oral dose of lemborexant-matched placebo tablet, on Day 1 of Treatment Periods 1, 2, or 3.
- Lemborexant 5 mg: Participants received a single oral dose of lemborexant 5 mg tablet, on Day 1 of Treatment Periods 1, 2, or 3.
- Lemborexant 10 mg: Participants received a single oral dose of lemborexant 10 mg tablet, on Day 1 of Treatment Periods 1, 2, or 3.
Arm/Group | Lemborexant-matched Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 68 | 69 | 68
minutes
  Baseline | 18.25 (2.621) | 18.28 (2.61) | 18.25 (2.621)
  Change at Day 2 After Each Treatment | -3.43 (4.424) | -4.56 (4.693) | -6.95 (4.967)
Statistical Analysis 1: Comparison: Lemborexant-matched Placebo vs Lemborexant 5 mg; Test type: Superiority or Other; p = 0.0262, Mixed Models Analysis — The mixed model included treatment, period and sequence as fixed effects, baseline (predose) measurement as a covariate, and participant nested within treatment sequence as a random effect; Mean Difference (Final Values) = -1.15, 95% CI 1-sided [lower limit -2.12]
Statistical Analysis 2: Comparison: Lemborexant-matched Placebo vs Lemborexant 10 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.48, 95% CI 1-sided [lower limit -4.46]

2. Secondary Outcome: Number of Participants With an Average SOL of Less Than (<) 8.0 Minutes for Each Treatment
Description: SOL is defined as the length of time that it takes to accomplish the transition from full wakefulness to sleep. The MSLT is a widely used method for objectively quantifying excessive, pathological, or pharmacologically induced residual sleepiness by measuring the number of minutes that it takes a participant to fall asleep. The MSLT was modified to include four SLTs, with the first starting at 45 minutes after morning wake time, and the subsequent three occurring at 30-minute intervals for a total of 4 SLT's per M-MSLT. Each SLT was scored to determine the latency in minutes (with precision to 0.5 minute) from lights off to sleep onset; trials during which sleep onset did not occur were assigned a latency of 20 minutes. The four SLTs for each participant were averaged to obtain the mean SOL.
Time Frame: Day 2 of each of three treatment periods that were separated by approximately 2 weeks (for a total of up to 6 weeks)
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose PD measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Flurazepam 30 mg: Participants received a single oral dose of flurazepam 30 mg capsule on Day 1 of Treatment Period 4.
Arm/Group | Lemborexant-matched Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
Number analyzed (Participants) | 68 | 69 | 68 | 68
Participants | 3 | 11 | 20 | 36
Statistical Analysis 1: Comparison: Lemborexant-matched Placebo vs Lemborexant 5 mg; Test type: Superiority or Other; p = 0.0215, McNemar — P-value was calculated based on non-missing two-way contingency table between placebo and study treatment
Statistical Analysis 2: Comparison: Lemborexant-matched Placebo vs Lemborexant 10 mg; Test type: Superiority or Other; p < 0.0001, McNemar — P-value was calculated based on non-missing two-way contingency table between placebo and study treatment
Statistical Analysis 3: Comparison: Lemborexant-matched Placebo vs Flurazepam 30 mg; Test type: Superiority or Other; p < 0.0001, McNemar — P-value was calculated based on non-missing two-way contingency table between placebo and study treatment

3. Secondary Outcome: Number of Participants Whose Treatment Difference (Under Either Dose of Lemborexant) Average SOL Score is More Than (>) 6.0 Minutes Shorter Than Placebo
Description: as for outcome 2
Time Frame: Day 2 of each of three treatment periods that are separated by approximately 2 weeks (for a total of up to 6 weeks)
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose PD measurement. Participants who were evaluable for this given measure at a given time point were included for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
Number analyzed (Participants) | 68 | 68 | 68
Participants | 9 | 20 | 35

4. Secondary Outcome: Number of Participants Whose Average SOL is <8.0 Minutes and >6.0 Minutes Shorter Than Placebo
Description: as for outcome 2
Time Frame: Day 2 of each of three treatment periods that are separated by approximately 2 weeks (for a total of up to 6 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
Number analyzed (Participants) | 68 | 68 | 68
Participants | 4 | 13 | 25

5. Secondary Outcome: Mean Change From Baseline in the Average SOL From the M-MSLT in Treatment Period 4
Description: as for outcome 2
Time Frame: Baseline, Day 2 of Treatment Period 4 (Week 6)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Flurazepam 30 mg
Number analyzed (Participants) | 68
minutes
  Baseline | 18.25 (2.621)
  Change at Day 2 of Treatment Period 4 | -9.49 (5.413)

6. Secondary Outcome: Mean Plasma Concentrations of Lemborexant and Metabolite M10 in the Morning Following M-MSLT
Description: The MSLT is a widely used method for objectively quantifying excessive, pathological, or pharmacologically induced residual sleepiness by measuring the number of minutes that it takes a participant to fall asleep. The MSLT was modified to include four SLTs, with the first starting at 45 minutes after morning wake time, and the subsequent three occurring at 30-minute intervals for a total of 4 SLT's per M-MSLT.
Time Frame: Days 2, 16 and 30 within 20 minutes after the end of 4th SLT (up to 155 minutes after wake time)
Population: The pharmacokinetic (PK) analysis set was the group of participants who received at least one dose of lemborexant and had at least one quantifiable postdose drug concentration. The PK analysis set where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 69 | 68
nanogram per milliliter (ng/mL)
  Lemborexant: Day 2: number analyzed (Participants) | 23 | 22
  Lemborexant: Day 2 | 2.285 (1.426) | 6.423 (3.262)
  Metabolite M10: Day 2: number analyzed (Participants) | 23 | 22
  Metabolite M10: Day 2 | 1.246 (0.792) | 2.582 (0.959)
  Lemborexant: Day 16: number analyzed (Participants) | 23 | 22
  Lemborexant: Day 16 | 3.236 (1.895) | 5.306 (3.175)
  Metabolite M10: Day 16: number analyzed (Participants) | 23 | 22
  Metabolite M10: Day 16 | 1.361 (0.634) | 2.689 (1.592)
  Lemborexant: Day 30: number analyzed (Participants) | 23 | 24
  Lemborexant: Day 30 | 2.020 (1.446) | 5.293 (4.293)
  Metabolite M10: Day 30: number analyzed (Participants) | 23 | 24
  Metabolite M10: Day 30 | 0.994 (0.639) | 2.304 (1.534)

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events (AEs) That Led to Death and Study Drug Discontinuation
Time Frame: From first dose of study drug up to Day 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant-matched Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
Number analyzed (Participants) | 68 | 69 | 68 | 68
Participants
  TEAEs | 2 | 5 | 8 | 5
  SAEs | 0 | 0 | 0 | 0
  AEs Leading to Death | 0 | 0 | 0 | 0
  AEs Leading to Discontinuation | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values
Time Frame: From first dose of study drug up to Day 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant-matched Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
Number analyzed (Participants) | 68 | 69 | 68 | 68
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs Values
Time Frame: From first dose of study drug up to Day 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant-matched Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
Number analyzed (Participants) | 68 | 69 | 68 | 68
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Shifts From Baseline in Electrocardiogram (ECG) Parameters
Time Frame: From first dose of study drug up to Day 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant-matched Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
Number analyzed (Participants) | 68 | 69 | 68 | 68
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Relationship Between PK Concentrations of Lemborexant and Sleepiness as Measured by M-MSLT
Description: Pearson correlation was used to calculate the relationship between PK concentration of lemborexant and sleepiness. The M-MSLT is a widely used method for objectively quantifying excessive, pathological, or pharmacologically induced residual sleepiness by measuring the number of minutes that it takes a participant to fall asleep. The MSLT was modified to include four SLTs, with the first starting at 45 minutes after morning wake time, and the subsequent three occurring at 30-minute intervals for a total of 4 SLT's per M-MSLT. Each SLT was scored to determine the latency in minutes (with precision to 0.5 minute) from lights off to sleep onset; trials during which sleep onset did not occur were assigned a latency of 20 minutes.
Time Frame: Baseline up to Day 44 (Week 6)
Population: The PK analysis set was the group of participants who received at least one dose of E2006 and had at least one quantifiable postdose drug concentration. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: correlation coefficient
Groups:
- Lemborexant 5 or 10 mg: All Participants: Participants received a single oral dose of lemborexant 5 mg or 10 mg tablet, on Day 1 of Treatment Periods 1, 2, or 3.
Arm/Group | Lemborexant 5 or 10 mg: All Participants
Number analyzed (Participants) | 62
correlation coefficient | -0.2746

ADVERSE EVENTS:
Time Frame: From date of first dose of study drug up to Day 54
Arm/Group | Lemborexant-matched Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Flurazepam 30 mg
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/69 | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69 | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 2/68 | 5/69 | 8/68 | 5/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lemborexant-matched Placebo (N=68) | Lemborexant 5 mg (N=69) | Lemborexant 10 mg (N=68) | Flurazepam 30 mg (N=68)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 3 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Hypnopompic hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes